CLINICAL TRIAL: NCT04931238
Title: Efficacy and Safety of a Recombinant Neutralizing Human Anti-SARS-CoV-2 Monoclonal Antibody JS016 in Chinese Hospitalized Patients With SARS-CoV-2 Infection (COVID-19): a Multicenter, Randomized, Open-label, Controlled Trial
Brief Title: Efficacy and Safety of JS016 in Patients With SARS-CoV-2 Infection (COVID-19)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Peking JS016
Record Dates: First submitted 2021-06-13; First posted 2021-06-18 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; JS016; spike (S) protein; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — etesevimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS016 treatment group (Experimental): Standard therapy + JS016 injection Standard therapy including vital sign monitoring, supplementary oxygen and respiratory support in accordance with the patient's oxygen saturation and respiratory condition.
  Interventions: Drug: JS016
- Control group (No Intervention): Standard therapy Standard therapy includes vital sign monitoring, supplementary oxygen and respiratory support in accordance with the patient's oxygen saturation and respiratory condition.

INTERVENTIONS:
Drug: JS016 — Single Intravenous Injection of JS016 with a dose of 50mg/kg
  Other Names: CB6-LALA
  Arms: JS016 treatment group

SUMMARY:
The human monoclonal antibody CB6 showed potent neutralization activity in vitro against SARS-CoV-2. CB6-LALA (also called JS016) has been developed for clinical use. Phase I trials among healthy volunteers has demonstrated a tolerable and safe drug profile of JS016. We aim to evaluate the efficacy and safety of JS016 in patients hospitalized with COVID-19.

DETAILED DESCRIPTION:
As the COVID-19 pandemic is emerging as a global healthcare crisis, scientists worldwide are actively developing prophylactic and therapeutic interventions. Neutralizing antibody therapies are being developed for the treatment of COVID-19. The human monoclonal antibody CB6 showed potent neutralization activity in vitro against SARS-CoV-2. The LALA mutation was introduced to the Fc portion of CB6 (CB6-LALA) to lower the risk of Fc-mediated acute lung injury in animals. CB6-LALA (also called JS016) has been developed for clinical use. Phase I trials among healthy volunteers has demonstrated a tolerable and safe drug profile of JS016. We aim to evaluate the efficacy and safety of JS016 in patients hospitalized with COVID-19. The data from this study will inform decisions of the clinical use of JS016.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute respiratory syndrome coronavirus2 (SARS-CoV-2) infection
* Within 7 days from the onset of clinical symptoms or 4 days from the onset of severe symptoms
* Consistent with the National Health Committee New Coronavirus pneumonia diagnosis and treatment plan (Eighth Edition), general or heavy diagnostic criteria.

Exclusion Criteria:

* Sever Covid-19 Infection patients
* SARS-Cov-2 specific antibodies (including IgM and IgG) were positive before included
* Cardiac function grade III or IV, or left ventricular ejection fraction < 30%
* History of known or suspected active pulmonary tuberculosis or extra-pulmonary tuberculosis
* Chronic renal failure needs maintenance dialysis
* History of solid malignant/tumor or hematological malignancy
* Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical status at 28 days | At 28 days from inclusion
  Clinical status at 28 days assessed using a six level ordinal scale，in this scale, 1 is the minimum score and presenting a better outcome as discharge, 2 means still in-hospital but no need of oxygen therapy, 3 presents in-hospital and needing of oxygen therapy, 4 presents in-hospital needing high flow nasal oxygen therapy or non-invasive mechanical ventilation, 5 presents in-hospital needing invasive mechanical ventilation or ECMO, 6 presents death and is the worse outcome as well.

SECONDARY OUTCOMES:
All cause mortality ascertained from data analysed to day 28 | At 28 days from inclusion
  All cause mortality ascertained from data analysed to day 28
Ventilator-free days within 28 days | At 28 days from inclusion
  Ventilator-free days within 28 days
Negative conversion rate of SARS-CoV-2 nucleic acid in on days 14 after randomization | At 14 days from inclusion
  Negative conversion rate of SARS-CoV-2 nucleic acid in on days 14 after
Average length of hospital stay | At 28 days from inclusion
  Average length of hospital stay

OTHER OUTCOMES:
The incidence Treatment-Emergent Adverse Events of JS016 | Everyday after inclusion up to 28 days from inclusion
  Incidence of Treatment-Emergent Adverse Events of JS016 includes the incidence of allergic reaction, secondary infection, liver dysfunction, acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Bin DU, Prof., Study Chair — Peking Union Medical College Hospital
Locations (4):
- China (4):
  - Li Weng, Beijing, Beijing Municipality
  - Shi Jiazhuang People's Hospital, Shijiazhuang, Hebei
  - The First Affliated Hospital of Harbin Medical University, Harbin, Hei Longjiang
  - Suihua first hospital, Suihua, Hei Longjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang L, Liu W, Yu X, Wu M, Reichert JM, Ho M. COVID-19 antibody therapeutics tracker: a global online database of antibody therapeutics for the prevention and treatment of COVID-19. Antib Ther. 2020 Jul;3(3):205-212. doi: 10.1093/abt/tbaa020. Epub 2020 Aug 19. PMID 33215063
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Dong R, Jiang L, Yang T, Wang C, Zhang Y, Chen X, Xie J, Guo Y, Weng L, Kang Y, Yu K, Qiu H, Du B; China Critical Care Clinical Trials Group (CCCCTG). Efficacy and Safety of SARS-CoV-2 Neutralizing Antibody JS016 in Hospitalized Chinese Patients with COVID-19: a Phase 2/3, Multicenter, Randomized, Open-Label, Controlled Trial. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0204521. doi: 10.1128/AAC.02045-21. Epub 2022 Mar 15. PMID 35191746